CLINICAL TRIAL: NCT06609850
Title: The Comparison of TACE-Lenvatinib With TACE-Lenvatinib-ablation for Intermediate Recurrent Hepatocellular Carcinoma: a Multicenter Randomized Control Study
Brief Title: The Comparison of TACE-Lenvatinib With TACE-Lenvatinib-ablation for Intermediate Recurrent Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 10
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Hepatocellular Carcinoma; Lenvatinib; Local Therapy; Ablation; Systemic Therapy
Keywords: Lenvatinb; Hepatocellular carcinoma; Microwave ablation; Radiofrequency ablation; Cryoablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE plus Lenvatinib (Active Comparator): TACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then a combination of lipiodol (5-15 ml), lobaplatin (30-50 mg), and Pirarubicin (30-50 mg) was infused into each tumor. We defined technical success as complete embolization of the tumor-feeding artery resulting in no tumor staining observed by angiogram at the end of procedure.
  Lenvatinb (12 mg (body weight ≥60 kg) , 8 mg (body weight <60 kg) orally once a day )
  Interventions: Procedure: TACE; Drug: Lenvatinb
- TACE plus Lenvatinib and ablation (Experimental): TACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then a combination of lipiodol (5-15 ml), lobaplatin (30-50 mg), and Pirarubicin (30-50 mg) was infused into each tumor. We defined technical success as complete embolization of the tumor-feeding artery resulting in no tumor staining observed by angiogram at the end of procedure.
  Lenvatinb (12 mg (body weight ≥60 kg) , 8 mg (body weight <60 kg) orally once a day ) Ablation (radiofrequency ablation, microwave ablation, cryoablation), ablation followed TACE within 6-8 weeks and Lenvatinib continued. Percutaneous ablation was performed by ultrasound or CT. The ablation success is evaluated by achieving an ablative margin of 0.5 cm or more than the tumor size.
  Interventions: Procedure: TACE; Procedure: Ablation; Drug: Lenvatinb

INTERVENTIONS:
Procedure: TACE — TACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then a combination of lipiodol (5-15 ml), lobaplatin (30-50 mg), and Pirarubicin (30-50 mg) was infused into each tumor. We defined technical success as complete embolization of the tumor-feeding artery resulting in no tumor staining observed by angiogram at the end of procedure.
Procedure: Ablation — Ablation (radiofrequency ablation, microwave ablation, cryoablation), ablation followed TACE within 6-8 weeks and Lenvatinib continued. Percutaneous ablation was performed by ultrasound or CT. The ablation success is evaluated by achieving an ablative margin of 0.5 cm or more than the tumor size.
  Arms: TACE plus Lenvatinib and ablation
Drug: Lenvatinb — Lenvatinb (12 mg (body weight ≥60 kg) , 8 mg (body weight <60 kg) orally once a day )

SUMMARY:
Studies have shown that combination therapy of TACE with Lenvatinib could achieve better survival outcomes than TACE alone for hepatocellular carcinoma (HCC) at BCLC B stage. However, whether patients could benefit from the ablation for intermediate recurrent HCC (RHCC) is still need high quality clinical evidence. This study is to evaluate the efficacy of ablation combined with TACE and Lenvatinib for the intermediate-stage RHCC.

DETAILED DESCRIPTION:
The evidence of ablation combined transarterial chemoembolisation (TACE) and Lenvatinib for intermediate-stage recurrent hepatocellular carcinoma (RHCC) is limited. Patient responses to this treatment vary because of the heterogeneous nature of RHCC. Thus, it is important to identify patients who are most likely to benefit from this three regimes therapy. The aim of this study is to comparison of TACE-Lenvatinib with TACE-Lenvatinib-ablation for intermediate RHCC.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years;
2. RHCC diagnosed by imaging;
3. intermediate-stage RHCC (two to three lesions which at least one was >3 cm in size or more than three tumors);
4. the tumor number was no more than six, and the maximum tumor diameter was ≤5 cm;
5. absence of extrahepatic metastasis or macrovascular invasion;
6. Child-Pugh class A or B;
7. TACE as initial treatment after tumor recurrence and showed no tumor progression after TACE.
8. life expectance >3 months;

Exclusion Criteria:

1. under 18 years or over 75 years of age;
2. primary intermediate-stage HCC;
3. RHCC with more than six tumors, or single RHCC

(5) RHCC >5cm; (6) extrahepatic metastasis; (7) macrovascular tumor thrombus;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 24 months
  PFS is defined as the time from the date of inclusion to the date of the first objectively documented tumor progression or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 36 month
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to mRECIST, is defined as partial response and complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, None Selected, China